CLINICAL TRIAL: NCT03571217
Title: The Cohort Study of Incidence and Disk Factors of Diabetic Retinopathy and Visual Impairment in Adults With Type 2 Diabetes
Brief Title: Shanghai Beixinjing Diabetic Eyes Study
Acronym: SBDES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Other Study IDs: YFZX2018003
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Diabetic Retinopathy; Visual Impairment; Diabetic Maculopathy
Keywords: Type 2 diabetes mellitus; diabetic retinopathy; visual impairment; diabetic choroidopathy
MeSH Terms: conditions — Diabetic Retinopathy; Vision Disorders; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic retinopathy cohort
- Mild visual impairment cohort

SUMMARY:
In industrialized nations diabetic retinopathy(DR) is the most frequent microvascular complication of type 2 diabetes mellitus and the leading cause of visual impairment and blindness in the working-age population. The well-accepted strategy for prevention and treatment of diabetic eye complications focused on confirmed diabetic retinopathy, diabetic macular edema, cataract, etc, and there was no definitive therapy for preclinical central visual acuity (CVA) impairment, mainly because of its unknown pathogenesis. In our previous population-based study, the prevalence rate of early CVA impairment was as high as 9.1%, and that obviously limits the effects of diabetic eye diseases prevention and early-stage treatment strategy. Of note, the choriocapillaris is the only route for metabolic exchange in the retina within the foveal avascular zone, it was speculated that early CVA impairment is related to diabetic choroidopathy (DC). Recent research shows that the decreased macular choriocapillaris vessel density (MCVD) in diabetic eye ,which indicating early ischemia, is already present before diabetic macular edema can be observed; we have observed subfoveal choroidal thickness (SFCT) decreased significantly in the early CVA impairment patients. However, up til now, there was no epidemiology report on early CVA impairment in Chinese diabetes population. In the present study, we plan to conduct a 10-year perspective cohort observation of 2217 Chinese type 2 diabetic residents without diabetic retinopathy, diabetic macular edema, cataract and other vision impairing diseases, trying to find out related physical and biochemical risk factors. The results will facilitate discriminating high risk groups of early CVA impairment in diabetic patients. In the same time, a quantitative relationship between SFCT change, MCVD change and CVA change will be established. This study will demonstrate the role of DC in the occurrence of preclinical CVA impairment, and provide important theoretic evidence of blocking agents which target on DC.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old;
* Diabetes mellitus (DM) was defined as either blood hemoglobin A1C≥6.5%, use of diabetic medication or a physician diagnosis of diabetes.

Exclusion Criteria:

* None;

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes mellitus. Diabetes mellitus (DM) was defined as either blood hemoglobin A1C≥6.5%, use of diabetic medication or a physician diagnosis of diabetes.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2014-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diabetic retinopathy | December 31，2024
  The DR grades are according to the well-accepted ''International Clinical Diabetic Retinopathy and Diabetic Macular Edema Disease Severity Scale''
mild visual impairment | December 31，2024
  Mild visual impairment was present if BCVA was < 20/25 but ≥ 20/63.
macular choriocapillaris vessel density(MCVD) | December 31，2024
  macular choriocapillaris vessel density
glycosylated hemoglobin | December 31，2024
  This test measures the average blood sugar control for the previous three months or so.
retinal thickness (RT) | December 31，2024
  Retinal thickness was defined as the distance from the internal limiting membrane to the interface of the photoreceptor outer segments and retinal pigment epithelium.
choroidal thickness (CT) | December 31，2024
  Choroidal thickness was measured from the outer border of the RPE to the inner border of the choroidoscleral interface.

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Zou, MD, PhD, Study Chair — Shanghai Eye Disease Prevention & Treatment Center
Locations (1):
- Shanghai Eye Disease Prevention & Treatment Center, Shanghai, Shanghai Municipality, China